CLINICAL TRIAL: NCT06906133
Title: Comparing Changes in Objective Measures of Sleep Quality During the Menstrual Cycle in Healthy Women: Association With Ovarian Hormones and Mood
Brief Title: Sleep Quality and the Menstrual Cycle
Status: Active, not recruiting | Type: Observational
Sponsor: University of Akureyri (Other)
Collaborators: Akureyri Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SQMCIceland
Record Dates: First submitted 2025-03-11; First posted 2025-04-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Sleep Quality
Keywords: Objectively measured sleep; Sleep quality; Sleep disorder breathing; Ovarian hormones; Mood; Menstrual cycle; Sleep duration
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 30 women with natural cycle: This pilot study will aim to recruit 60 women (18-40 years) to participate; 30 natural menstrual cycle/30 that use hormonal contraceptives.
  Interventions: Other: Urinary-hCG
- 30 women using hormonal contraceptives: This pilot study will aim to recruit 60 women (18-40 years) to participate; 30 natural menstrual cycle/30 that use hormonal contraceptives.
  Interventions: Other: Urinary-hCG

INTERVENTIONS:
Other: Urinary-hCG — Ovulation days will be detected using a commercial urine test for luteinizing hormone (LH) (PREGMATE, Ovulation Midstream Test Predictor Kit; sensitivity level:25mlU/mL). Participants will be instructed to use ovulation tests, starting 5 days before the expected ovulation (day 10) and for the next 7-10 days or until the first the first positive results are detected notify the study co-ordinator and share a photo of the results. Then participants will be asked to continue using the ovulation test for 3 more days.

SUMMARY:
This study aims to examine how ovarian hormone fluctuations across the menstrual cycle affect sleep patterns. Using objective sleep tracking, hormone phase assessment, and validated questionnaires, it will assess changes in sleep quality, duration, menstrual symptoms, sleepiness, chronotype, anxiety, and depression over one full cycle.

DETAILED DESCRIPTION:
Study design:

A prospective community-based study focusing on women of reproductive age (18-36 years) designed to evaluate whether the phase of the menstrual cycle affects sleep quality and/or sleep duration. The study methods and results will be reported following the Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) for cross-sectional studies.

Recruitment of Participants:

If approved by the local research ethics committee (VSN-2411037), the study will be registered at ClinicalTrials.gov and women of reproductive age (18-36 years) will be recruited. The main method of recruitment will be a message sent through social media messaging system. Women residing in Iceland will be invited to participate. All the women participating in the study will be provided with information about the study and asked to sign a written informed consent before entering the study. All participants will be allowed to withdraw from the study at any time. Participants will not be financially compensated for their participation.

General Health & Sleep Evaluation (subjective):

Before starting the program, women that have signed an informed consent to participate will attend an introductory meeting (approximately 30 minutes), for women not living in Akureyri and neighbourhood but want to participate in the study meeting will be held virtually. Women still interested to participate after the meeting be asked to fill out questionnaires to evaluate:

1. Demographics and general health.
2. The impact of menstrual distress and its impact on psychological well-being. The Menstrual Distress Questionnaire (MEDI-Q) is a twenty-five-item questionnaire with reliability of 0.84 and score >=20 indicating menstruation-related distress.
3. Level of daytime sleepiness. The Epworth sleepiness scale (ESS), is an eight-item questionnaire with reliability 0.73 and score of 11-15 indicating mild-moderate sleepiness and >=16 severe sleepiness.
4. Nighttime and daytime components of insomnia. The Insomnia severity index (ISI), is a seven-item questionnaire with reliability 0.83 and score of 15-21 indicating mild-moderate and >=22 severe insomnia symptoms.
5. Severity of anxiety. The General anxiety disorder-7 scale (GAD-7), a seven-item questionnaire with reliability 0.91 and score of 10-14 indicating mild-moderate and >=15 severe anxiety symptoms.
6. Severity of depression. The Beck's depression inventory-II (BDI-II), is a ten-item questionnaire with reliability 0.90 and score of 20-28 indicating moderate and >=29 severe depression symptoms.
7. Preferred timing of sleep and activity. The Morningness-Eveningness questionnaire (MEQ), is a nineteen-item questionnaire with reliability 0.68 and scores of 16-41 indicating evening type, 42-58 intermediate type and 59-86 morning type.
8. Preferred food choices.

Menstrual Cycle Tracking:

Ovulation days will be detected using a commercial urine test for luteinizing hormone (LH) (PREGMATE, Ovulation Midstream Test Predictor Kit; sensitivity level:25mlU/mL). Participants will be instructed to use ovulation tests, starting 5 days before the expected ovulation (day 10) and for the next 7-10 days or until the first the first positive results are detected notify the study co-ordinator and share a photo of the results. Then participants will be asked to continue using the ovulation test for 3 more days.

Sleep Evaluation (Objective):

Participants will asked to record their sleep for all nights over period of one-menstrual cycle (starting the first day of their period and ending when the next period starts) with FDA_cleared_182618 home sleep test (HST) (SleepImage System; MyCardio LLC, Denver, Colorado, US). This test also complies with the EU Medical Device Regulation (CE mark 2862).

The SleepImage System comprises a finger-worn data-collection device including a photoplethysmography sensor (PPG) and a mobile application that sends the data to a secure cloud-based portal for data analysis (Figure 1). The data-recorder collects plethysmography-signal (PLETH) and oxygen saturation (SpO2) information that is automatically analyzed utilizing cardiopulmonary-coupling (CPC) algorithms to derive sleep information, then combined with SpO2 to calculate apnea hypopnea index (AHI). The CPC-method has been described in detail in several prior publications. In brief, the method is based on recording and analyzing dynamics in signals controlled by the autonomic nervous system (ANS) during sleep, more specifically by calculating the coherence between heart/pulse rate variability and respiratory excursions derived from a PLETH-signal. Then, a spectral analysis is performed to generate sleep stages. Non-rapid eye movement (NREM) sleep is presented as bimodal: stable sleep (high-frequency coupling, HFC;0.1-0.5Hz) that includes all electro-encephalogram (EEG) estimated NREM-3 and part of NREM-2 sleep, and is associated with periods of stable breathing, non-cyclic alternating pattern (CAP) EEG, increased delta power and blood pressure dipping and unstable-sleep (low-frequency coupling, LFC;0.01-0.1Hz) that includes all NREM-1 and portion of NREM-2 associated with sleep instability, characterized by variability of tidal volumes, blood pressure non-dipping and CAP-EEG. Wake and rapid eye movement (REM) sleep show very low-frequency coupling characteristics (vLFC;0-0.01Hz). The output includes sleep onset (SO), sleep conclusion (SC), sleep duration, total sleep time (TST), wake after sleep onset (WASO), sleep efficiency (SE), sleep quality index (SQI) displayed on a scale of 0-100, and AHI.

Investigators have in a previous study confirmed the feasibility to use this method for multi-night testing.

ELIGIBILITY:
Inclusion Criteria:

1. Women, 18-36 years
2. Body Mass Index (BMI) <=35
3. Regular menstrual cycle, defined as: length of menstrual cycle 22-35 days and length of menses <10 days.
4. Women with natural menstrual cycle (i.e., do not use any type of hormonal contraceptives) and women using contraceptives (comparison group).

Exclusion Criteria:

Previously diagnosed with:

1. Sleep apnea, clinical insomnia, restless leg syndrome, narcolepsy.
2. Shift work and trans-meridian travel during the study period.
3. Chronic atrial fibrillation or ventricular trigemini, severe uncontrolled asthma, or other pulmonary diseases.
4. Premenstrual Dysphoric Disorder (PMDD) or severe Premenstrual Syndrome (PMS).
5. Other severe medical conditions that may affect cerebral metabolism, cancer, diabetes, rheumatoid arthritis, or other chronic health conditions.
6. Severe psychiatric conditions, Major Depressive disorder, Generalized Anxiety Disorder, Bipolar Disorder, Personality Disorder, OCD, Schizophrenia.
7. Severe neurological conditions, epilepsy, traumatic brain injury, and previous neurosurgery.
8. Habitual smokers and other habitual substance abuse or dependence on substances.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: This pilot study will aim to recruit 60 women (18-36 years) to participate; 30 natural menstrual cycle/30 that use hormonal contraceptives.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Sleep duration | From March 15 2025 to January 15 2026
  1. Sleep duration - calculated in hours. minutes.
  Sleep output is measured utilizing home sleep test (SleepImage) that is FDA cleared and EU Medical Device Regulation (CE marked) compliant sleep test calculating:
  Sleep Duration (SD) based on calculating the time from sleep onset (SO) to sleep conclusion (SC) in hours and minutes.
Sleep quality | From March 15 2025 to January 15 2026
  2. Sleep Quality - based on sleep quality index (SQI) on a scale of 0-100.
  Sleep output is measured utilizing home sleep test (SleepImage) that is FDA cleared and EU Medical Device Regulation (CE marked) compliant sleep test calculating: Sleep Quality Index (SQI) is summary index of all sleep parameters presented on a scale of 0-100.

SECONDARY OUTCOMES:
Ovulation days | From March 15 2025 to January 15 2026
  1. Ovulation days will be detected utilizing ovulation midstream test predictor kit reporting results as positive or negative.
  Ovulation days will be detected using a commercial urine test for luteinizing hormone (LH) (PREGMATE, Ovulation Midstream Test Predictor Kit; sensitivity level:25mlU/mL). Participants will be instructed to use ovulation tests, starting 5 days before the expected ovulation (day 10) and for the next 7-10 days or until the first the first positive results are detected notify the study co-ordinator and share a photo of the results. Then participants will be asked to continue using the ovulation test for 3 more days.

CONTACTS AND LOCATIONS:
Overall Officials: Sólveig Magnúsdóttir, MD, MSc, MBA., Principal Investigator — MyCardio
Locations (2):
- Iceland (2):
  - Akureyri Hospital, Akureyri
  - University of Akureyri, Akureyri

IPD SHARING:
Plan to Share IPD: Undecided
The data collected during this study is not publicly available due to General Data Protection Regulations (GDPR) reasons.

REFERENCES:
- [Background] Lu M, Penzel T, Thomas RJ. Cardiopulmonary Coupling. Adv Exp Med Biol. 2022;1384:185-204. doi: 10.1007/978-3-031-06413-5_11. PMID 36217085
- [Background] Chung KF, Kan KK, Yeung WF. Assessing insomnia in adolescents: comparison of Insomnia Severity Index, Athens Insomnia Scale and Sleep Quality Index. Sleep Med. 2011 May;12(5):463-70. doi: 10.1016/j.sleep.2010.09.019. Epub 2011 Apr 13. PMID 21493134
- [Background] Cassioli E, Rossi E, Melani G, Faldi M, Rellini AH, Wyatt RB, Oester C, Vannuccini S, Petraglia F, Ricca V, Castellini G. The menstrual distress questionnaire (MEDI-Q): reliability and validity of the English version. Gynecol Endocrinol. 2023 Jun 19;39(1):2227275. doi: 10.1080/09513590.2023.2227275. PMID 37356456
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Alzueta E, de Zambotti M, Javitz H, Dulai T, Albinni B, Simon KC, Sattari N, Zhang J, Shuster A, Mednick SC, Baker FC. Tracking Sleep, Temperature, Heart Rate, and Daily Symptoms Across the Menstrual Cycle with the Oura Ring in Healthy Women. Int J Womens Health. 2022 Apr 8;14:491-503. doi: 10.2147/IJWH.S341917. eCollection 2022. PMID 35422659
- [Background] Li DX, Romans S, De Souza MJ, Murray B, Einstein G. Actigraphic and self-reported sleep quality in women: associations with ovarian hormones and mood. Sleep Med. 2015 Oct;16(10):1217-24. doi: 10.1016/j.sleep.2015.06.009. Epub 2015 Jun 26. PMID 26429749
- [Background] Pengo MF, Won CH, Bourjeily G. Sleep in Women Across the Life Span. Chest. 2018 Jul;154(1):196-206. doi: 10.1016/j.chest.2018.04.005. Epub 2018 Apr 19. PMID 29679598
- Available data/document: Information site for participants (in Icelandic) — https://www.unak.is/is/rannsoknir/rannsoknir-vid-ha/svefn